CLINICAL TRIAL: NCT02204683
Title: A Pharmacokinetic Study of Intravitreal Aflibercept Injection in Vitrectomized and Non-vitrectomized Eyes With Wet Age-related Macular Degeneration (the DRAW Study)
Brief Title: Pharmacokinetic Study of Intravitreal Aflibercept Injection in Eyes With Wet Age-related Macular Degeneration
Acronym: DRAW
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0334-14-FB
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Neovascular Macular Degeneration
Keywords: AMD; Neovascularization; macular degeneration; wet macular degeneration; vitrectomy
MeSH Terms: conditions — Neovascularization, Pathologic; Macular Degeneration; Wet Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aflibercept (Other): Subjects who have had a vitrectomy previously
  Interventions: Drug: Aflibercept
- Aflibercept in Non-Vitrectomized eyes (Other): Patients who have not had vitrectomy.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Intravitreal aflibercept
  Other Names: Eylea

SUMMARY:
The main goal is to study way that aflibercept injection behaves in the eye and in the body of patients with wet macular degeneration, in patients who have had previous vitreous removal surgery.

DETAILED DESCRIPTION:
A pharmacokinetic study of intravitreal Aflibercept injection vitrectomized and non-vitrectomized eyes with Wet age-related macular degeneration (the DRAW study).

The primary objective is to investigate and characterize the intraocular pharmacokinetics of intravitreal aflibercept injection in vitrectomized and non-vitrectomized eyes with neovascular Age-related Macular Degeneration (AMD). The secondary objective is to assess the systemic pharmacokinetics of intravitreal aflibercept injection.

Little information is known about the intraocular pharmacokinetics of intravitreal aflibercept injection in human eyes. In addition, the durability of intravitreal aflibercept injection in vitrectomized eyes is not known, since individuals with a history of vitrectomy have been excluded from clinical trials in neovascular AMD. There have also been no studies on systemic levels following intravitreal aflibercept injection, which would have implications for normal vascular hemostasis and wound repair in which vascular endothelial growth factor (VEGF) plays an important role. The proposed research will fill in these gaps in the knowledge base for intravitreal aflibercept injection.

Two arms (non-vitrectomized, and vitrectomized) are included in the study to evaluate the intraocular and systemic pharmacokinetics of intravitreal aflibercept injection The study involves neovascular AMD patients divided into two groups: 5 patients with history of vitrectomy and 10 patients with no history of vitrectomy. Plasma blood and aqueous fluid will be collected at baseline, then 2mg of intravitreal aflibercept injection administered at time 0 (day 0). At 4 hours post injection, plasma (blood) and aqueous fluid will be collected again, as well as on days 1, 3, 7,14, and 28. Intravitreal aflibercept injection levels in the samples will be assessed and compared among the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 50 years
2. Active neovascular AMD, with no history of treatment in the study eye 2.1 10 patients with non-vitrectomized eyes 2.2 5 patients with vitrectomized eyes
3. Phakic and pseudophakic eyes are allowed in the study.
4. Willing and able to provide written informed consent after the nature of the study has been explained, and prior to any research-related procedures
5. Willing and able to comply with clinic visits and study-related procedures

Exclusion Criteria:

1. Presence of other retinal vascular diseases (diabetic retinopathy, vein occlusion) that could affect the VEGF levels within the eye
2. Known hypersensitivity to aflibercept
3. Autoimmune disease of the anterior segment or posterior chamber including chronic keratoconjunctivitis sicca, uveitis, iritis/scleritis, blepharitis of either eye
4. Infectious conjunctivitis, keratitis, or endophthalmitis of either eye
5. Previous participation in any studies of investigational drugs within 1 month preceding Day 0
6. Any clinically significant acute or chronic medical condition that would preclude participation in a clinical study
7. Pregnant or breast-feeding women
8. Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device (IUD); bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly) *Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-09-05 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2016-12-14 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) aflibercept aqueous | 28 days
  The primary endpoint in the study consists of intraocular aflibercept (free and bound) concentrations following intravitreal aflibercept injection.

SECONDARY OUTCOMES:
PK Aflibercept plasma | 28 days
  The secondary endpoints are plasma concentrations of aflibercept (free and bound) following intravitreal aflibercept injection.

CONTACTS AND LOCATIONS:
Overall Officials: Diana V Do, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Truhlsen Eye Institute, Omaha, Nebraska, United States